CLINICAL TRIAL: NCT03549481
Title: Role of TIMI, PURSUIT and GRACE Risk Scores in Predicting LV Remodeling in Patients With Acute Coronary Syndrome
Brief Title: Predictive Value of Risk Scores in Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: shaimaa Mostafa (Other)
Responsible Party: Sponsor-Investigator, shaimaa Mostafa, assistant professor of cardiovascular medicicne, Benha University
Organization: Benha University (Other)
Other Study IDs: 3 SH research
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Acute Coronary Syndrome; Left Ventricle Remodeling; Risk Scores
Keywords: risk score; acute coronary syndrome; left ventricular remodelng
MeSH Terms: conditions — Acute Coronary Syndrome; Ventricular Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
role of different risk scores in acute coronary syndrome to predict left ventricular remodeling

DETAILED DESCRIPTION:
patients with acute coronary syndrome (STEMI, NSTEMI, UA) will be included and different risk scores will be calculated for each patient.

after that in-hospital and short-term outcome beside left ventricular systolic and diastolic functions (at admission and 3m later) will be assessed to be correlated with different risk scores to determine which score system was able to predict left ventricular remodeling and what was the cut off value, sensitivity, and specificity of the score

ELIGIBILITY:
Inclusion Criteria:

* patients with acute coronary syndrome

Exclusion Criteria:

* previous acute coronary syndrome previous PCI or CABG chronic renal disease decompensated liver disease patient refusal to participate patients dropped during follow up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients of both gender with acute coronary syndrome
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
left ventricular remodeling | 3 months
  end diastolic volume, end systolic volume, ejection fraction
in hospital and short term outcme | 3 months
  re-infarction, death, arrhythmia

CONTACTS AND LOCATIONS:
Locations (1):
- shaimaa Mostafa, Cairo, Egypt